CLINICAL TRIAL: NCT05567978
Title: Evaluation of the Correlation Between the 2 Pupillometry Indexes (QPI and NPI) in Cerebral Palsy Patients
Brief Title: Comparison of 2 Pupillometric Indices in Cerebral Brain Patients
Acronym: LYNX
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital Brussel (Unknown); Ramon y Cajal University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0245
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pupillometry Index in Brain Lesion
Keywords: Brain lesion; pupillometry index; neurological outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: pupillometry index — Admission to the intensive care unit, measurement of pupillometry index every 4 hours for 7 days or at extubation of brain damaged patients

SUMMARY:
Pupillary examination, and in particular pupillary reactivity to light, is fundamental to the monitoring and follow-up in intensive care units of patients with acute brain injury. A pupillometric index combining different parameters of pupillary light reflex has been described as predictive of intracranial hypertension and the neurological outcome of the patient.

DETAILED DESCRIPTION:
Pupillary examination, and in particular pupillary reactivity to light, is fundamental for the monitoring and follow-up in intensive care units of patients with acute brain injury. Intracranial pressure monitoring and pupillometry measurement are thus part of the routine practice of intensive care unit management of brain injured patients. Furthermore, elevated intracranial pressure in brain injured patients admitted to the ICU is associated with a poor prognosis, and very high intracranial pressure is a life-threatening situation.

A pupillometry index combining different parameters of pupillary light reflex has been described as having predictive value of intracranial hypertension and neurological outcome of the patient: the "NPi". Another manufacturer IdMed, Marseille, France proposes an index: the QPI (Quantitative Pupillometry Index), based on a statistical classification of the amplitude of the light reflex.

The aim of this study is to show that :

* QPI is equivalent to NPI
* An abnormal value of the pupillometry indexes (NPI/QPI) is predictive of high intracranial pressure.
* An abnormal value of pupillometry indexes (NPI/QPI) is predictive of a poor neurological outcome at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients admitted for any brain injury: traumatic, intracranial hemorrhage, subarachnoid hemorrhage
* Pupillometry available as a standard assessment tool.
* Patient intubated/ventilated for neurological reasons for more than 12 hours

Exclusion Criteria:

* Non-intensive care patients
* Facial and or ocular trauma not allowing pupillometry evaluation
* Patients admitted to the ICU with a life expectancy of < 24 hours
* Protected persons (under guardianship, curators, pregnant or breastfeeding women, persons deprived of liberty, persons not subject to a psychiatric measure)
* Patients not affiliated to a social security system
* Patients who object to the use of their data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient admitted for a traumatic brain injury, intracranial hemorrhage, or subarachnoid hemorrhage and for whom a pupillometry indication is retained
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the correlation of the 2 existing NPI pupillometry index ans the IPQ in cerebral palsy patients | at 7 days
  The NPI and QPI value between 0 and 5

SECONDARY OUTCOMES:
To assess the relationship between pupillometry indices (NPI/QPI) and intracranial hypertension | at 7 days
  number of intracranial hypertension based on ICP value >5mns
To evaluate the contribution of the QPI and NPI indexes in predicting mortality and neurological outcome compared to existing scores (IMPACT, CRASH) | 6 months
  GOS-E at 6 months
Describe the satisfaction of the caregivers on the use of these 2 pupillometry devices | at 1 year
  Satisfaction questionnaire for users ( not at all satisfied, moderately satisfied, very satisfied) scale from 0 to 100. 100 is the best score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble ALPES, Grenoble, France, France

IPD SHARING:
Plan to Share IPD: No
Because of the observational/exploratory nature of the study, no formal sample size calculation has been performed. However, it is planned to recruit a total of at least 30 patients (traumatic brain injury, intracranial hemorrhage, subarachnoid hemorrhage), over a 12-month period.
  Data will be described in numbers and percentages for qualitative data, and in quartiles and means/standard deviation for quantitative characteristics.

REFERENCES:
- [Background] Sharshar T, Citerio G, Andrews PJ, Chieregato A, Latronico N, Menon DK, Puybasset L, Sandroni C, Stevens RD. Neurological examination of critically ill patients: a pragmatic approach. Report of an ESICM expert panel. Intensive Care Med. 2014 Apr;40(4):484-95. doi: 10.1007/s00134-014-3214-y. Epub 2014 Feb 13. PMID 24522878
- [Background] Chen JW, Gombart ZJ, Rogers S, Gardiner SK, Cecil S, Bullock RM. Pupillary reactivity as an early indicator of increased intracranial pressure: The introduction of the Neurological Pupil index. Surg Neurol Int. 2011;2:82. doi: 10.4103/2152-7806.82248. Epub 2011 Jun 21. PMID 21748035
- [Background] Chen JW, Vakil-Gilani K, Williamson KL, Cecil S. Infrared pupillometry, the Neurological Pupil index and unilateral pupillary dilation after traumatic brain injury: implications for treatment paradigms. Springerplus. 2014 Sep 23;3:548. doi: 10.1186/2193-1801-3-548. eCollection 2014. PMID 25332854
- [Background] Larson MD, Behrends M. Portable infrared pupillometry: a review. Anesth Analg. 2015 Jun;120(6):1242-53. doi: 10.1213/ANE.0000000000000314. PMID 25988634
- [Background] Larson MD, Singh V. Portable infrared pupillometry in critical care. Crit Care. 2016 Jun 22;20(1):161. doi: 10.1186/s13054-016-1349-7. PMID 27329287
- [Background] Volpi PC, Robba C, Rota M, Vargiolu A, Citerio G. Trajectories of early secondary insults correlate to outcomes of traumatic brain injury: results from a large, single centre, observational study. BMC Emerg Med. 2018 Dec 5;18(1):52. doi: 10.1186/s12873-018-0197-y. PMID 30518336
- [Background] Han J, King NK, Neilson SJ, Gandhi MP, Ng I. External validation of the CRASH and IMPACT prognostic models in severe traumatic brain injury. J Neurotrauma. 2014 Jul 1;31(13):1146-52. doi: 10.1089/neu.2013.3003. Epub 2014 May 12. PMID 24568201
- [Background] Couret D, Boumaza D, Grisotto C, Triglia T, Pellegrini L, Ocquidant P, Bruder NJ, Velly LJ. Reliability of standard pupillometry practice in neurocritical care: an observational, double-blinded study. Crit Care. 2016 Mar 13;20:99. doi: 10.1186/s13054-016-1239-z. PMID 27072310
- [Background] Couret D, Simeone P, Freppel S, Velly L. The effect of ambient-light conditions on quantitative pupillometry: a history of rubber cup. Neurocrit Care. 2019 Apr;30(2):492-493. doi: 10.1007/s12028-018-0664-z. No abstract available. PMID 30604030
- [Background] Olson DM, Stutzman S, Saju C, Wilson M, Zhao W, Aiyagari V. Interrater Reliability of Pupillary Assessments. Neurocrit Care. 2016 Apr;24(2):251-7. doi: 10.1007/s12028-015-0182-1. PMID 26381281